CLINICAL TRIAL: NCT01727596
Title: The Effects and Predictors of Patella Taping in the Treatment of Patellafemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 200904034R
Record Dates: First submitted 2009-12-18; First posted 2012-11-16 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Other: taping

INTERVENTIONS:
Other: taping — Briefly, the patella was manually displaced medially, and maintained in the position by Tex Tape (Kinesio Holding Corporation, Albuquerque, NM)
  Other Names: McConnell taping, patella tapping

SUMMARY:
Background: Taping has been used for more than 20 years for patellofemoral pain syndrome (PFPS) but the effectiveness is still controversial.

Purpose: This prospective study was conducted to investigate the effect and predictors of effectiveness of taping in treating PFPS.

Study design: Prospective cohort study Methods: One hundred consecutive patients with the diagnosis of PFPS were included in the study. Factors including sex, age, body mass index (BMI), Q angle, lateral patella displacement (LPD), lateral patellofemoral angle (LPA) and pre-taping pain score were measured. One well-trained therapist applied adhesive tape to each patient by McConnell approach. Before and after taping, patients completed a visual analog pain scale (VAS) after performing a step-down from an 8-inch platform. Paired-t test was used for the difference of the VAS score measured before and after taping. Patients with improvement of more than 1 point in VAS score after taping were considered responsible, and others were non-responsible. The results were analyzed by logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* (1) between the age of 20 to 60 years, (2) antero-, retro-, or peri-patellar pain from at least two of the following: prolonged sitting, ascending or descending stairs, prolonged walking, squatting, and (3) insidious onset of symptoms unrelated to a traumatic incident.

Exclusion Criteria:

* (1) symptoms or signs of any intrarticular derangement of the knee joint, such as effusion, ligament laxity, and meniscal tear, (2) tenderness over the patella tendon, iliotibial band, or pes anserinus tendons, (3) Osgood-Schlatter disease or Sinding-Larsen-Joahanssen syndromes, (4) referral pain from hip or lumbar region, (5) a history of patellar dislocation, previous knee surgery or infection, (6) malignancy, (7) present pregnancy, (8) recent treatment for the PFPS, such as physiotherapy, non-steroid anti-inflammatory or corticosteroid medication, (9) advanced osteoarthritis of the knee joint.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
VAS score | two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Chuan Jiang, M.D. PHD, Study Chair — National Taiwan University Hospital
Locations (1):
- NTUH, Taipei, Taiwan